CLINICAL TRIAL: NCT04924855
Title: Estimation of Dynamics of Humoral Immunity in COVID-19 Vaccined Health Care Workers
Brief Title: Immunity After COVID-19 Vaccination
Acronym: IACOVV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Sponsor
Other Study IDs: UR17DN05-3
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Tunis Military Hospital Staff Vaccinated Against Covid 19
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood sampling (4 per year)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling (4 per year) — Blood sampling (4 per year)

SUMMARY:
The purpose of the research is to evaluate kinetic after vaccination to the COVID-19 coronavirus by measurements of specific and neutralizant antibodies for spike antigenic sequences .

This work will allow us to follow the efficacy and tolerance of the vaccine over a year, to evaluate the antibody profile, their kinetics, the fraction of neutralising antibodies and will also allow us to understand the attitudes to be taken to ensure the best protection for our staff

DETAILED DESCRIPTION:
Our objective is to follow the hospital staff after vaccination, for this we will include two groups of participants:

G1: vaccinated staff who did not contract the virus (at the date of vaccination) and who had a serology <0 at least at D7 of the date of vaccination dose 1 (known serological value) G2: vaccinated personnel who have contracted the virus with a PCR + and who have positive serology at least at D7 of the date of vaccination (known serological value)

ELIGIBILITY:
Inclusion Criteria:

RB-approved informed consent, age 18 years or older, male or female, anyone considering COVID-19 vaccination or anyone that has received COVID-19 vaccination.

Subjects can enroll at anytime after vaccination even though they may not have enrolled before vaccination.

Sampling Frequency and timing: Up to 8 total samples in 12 months -

Exclusion Criteria:

Exclusion: Failure to provide informed consent

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: military health personnel vaccinated at tunis military hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Vaccine effectiveness | 1 year
  Vaccine effectiveness as measured by the number of positive PCRs in one year
Vaccine effectiveness | 1 year
  antibody kinetics

SECONDARY OUTCOMES:
the tolerance of the vaccine | 1 year
  post-vaccination adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- HMPIT vaccination committee, Tunis, Please Select..., Tunisia

IPD SHARING:
Plan to Share IPD: No